CLINICAL TRIAL: NCT01821820
Title: Influence of Pistachios on Performance and Exercise-induced Inflammation, Oxidative Stress, and Immune Dysfunction in Athletes: a Metabolomics-based Approach.
Brief Title: Pistachios, Performance, Metabolomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 13-0064
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Inflammation; Oxidative Stress; Immune Dysfunction
Keywords: Inflammation; Oxidative stress; Immune dysfunction; Metabolites
MeSH Terms: conditions — Inflammation; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pistachios (Experimental): Pistachio treatment (3 oz/d) for two weeks; 3 oz pistachio nuts and water (1.5 oz. before, and 1.5 oz during) cycling 75 km.
  Interventions: Other: Pistachios
- No pistachios (No Intervention): No pistachios for two weeks, or before and during 75 km cycling.

INTERVENTIONS:
Other: Pistachios
  Arms: Pistachios

SUMMARY:
Ingestion of 3 ounces of pistachio nuts per day for two weeks before and the day of cycling intensely for 75 kilometers will support substrate utilization during exercise (as determined through metabolomics) and improve performance compared to water only, and attenuate inflammation, oxidative stress, and immune dysfunction during 24 hours of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male endurance cyclists
* Capable of exercising for 2.5 h at a high intensity in the lab
* Ages 18-55
* Agree to train normally and stay weight stable.
* Agree to avoid the use of large dose vitamin/mineral supplements
* Agree to avoid herbs and medications that influence inflammation

Exclusion Criteria:

* Regularly take supplements or medicines known to effect inflammation.
* At moderate or high risk for cardiovascular disease.
* Younger than 18 or older than 55 years of age.
* No history of competing in cycling races.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Shifts in metabolites (metabolomics) | 14-day period
  Shifts in metabolites pre-and post-14-days supplementation, and then after 75-km cycling, and the next morning.

SECONDARY OUTCOMES:
Inflammation | 14-day period
  Pre- and post-14 d supplementation, and following 75-km cycling; plasma IL-6, IL-8, IL-10, TNF-alpha, G-CSF, MCP-1; C-reactive protein
Immune Function | 14-day period
  Pre- and post-14 days supplementation, and following 75-km cycling; granulocyte and monocyte phagocytosis and oxidative burst activity; leukoycte differential
Oxidative Stress | 14-day period
  Pre- and post-14 days supplementation, and following 75-km cycling; RBC glutathione, protein carbonyls, ORAC, FRAP, F2-isoprostanes

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- ASU Human Performance Laboratory, North Carolina Research Campus, Kannapolis, North Carolina, United States

REFERENCES:
- [Background] Dreher ML. Pistachio nuts: composition and potential health benefits. Nutr Rev. 2012 Apr;70(4):234-40. doi: 10.1111/j.1753-4887.2011.00467.x. PMID 22458696
- [Derived] Nieman DC, Scherr J, Luo B, Meaney MP, Dreau D, Sha W, Dew DA, Henson DA, Pappan KL. Influence of pistachios on performance and exercise-induced inflammation, oxidative stress, immune dysfunction, and metabolite shifts in cyclists: a randomized, crossover trial. PLoS One. 2014 Nov 19;9(11):e113725. doi: 10.1371/journal.pone.0113725. eCollection 2014. PMID 25409020
- See also: Lab web site — http://www.ncrc.appstate.edu